CLINICAL TRIAL: NCT01539434
Title: Behavioral Medicine Intervention to Maintain Physical Capacity and Level of Physical Activity in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Behavioral Intervention to Maintain Physical Capacity and Activity in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOU-2012-MEKW
Record Dates: First submitted 2012-02-08; First posted 2012-02-27 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Behavioral intervention; Physical capacity; Physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioural intervention (Experimental): Patients in the behavioural intervention group will get a personal meeting with the physiotherapist and get advice about the value of physical activity and also get recommendations on how to be physically active. The behavioural intervention to support physical activity behaviour includes weekly motivational interviewing telephone calls for the first month, two telephone calls for the following two months and thereafter monthly telephone calls.
  Interventions: Behavioral: Behavioural intervention
- Usual care group (Active Comparator): Patients in the usual care group will get a personal meeting with the physiotherapist and get advice about the value of physical activity and also get recommendations on how to be physically active.
  Interventions: Behavioral: Usual care group

INTERVENTIONS:
Behavioral: Behavioural intervention — Patients in the behavioural intervention group will get a personal meeting with the physiotherapist and get advice about the value of physical activity and also get recommendations on how to be physically active. The behavioural intervention to support physical activity behaviour includes weekly motivational interviewing telephone calls for the first month, two telephone calls for the following two months and thereafter monthly telephone calls.
  Other Names: Physical capacity; Physical activity
  Arms: Behavioural intervention
Behavioral: Usual care group — Patients in the usual care group will get a personal meeting with the physiotherapist and get advice about the value of physical activity and also get recommendations on how to be physically active.
  Other Names: Physical capacity; Physical activity
  Arms: Usual care group

SUMMARY:
The purpose of this study is to investigate to what extent patients with COPD, who have participated in physical training for 12 weeks, can maintain their physical activity behaviour and physical capacity on a long-term basis if they get a behavioural medicine intervention.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive disease and the number of patients is increasing. Persons with COPD have a low physical capacity and a low physical activity level. The risk of premature morbidity and mortality is high especially in persons with a low level of physical capacity and activity. Rehabilitation including physical training is recommended and results in decreased morbidity and mortality and increased physical capacity and quality of life. Unfortunately improvements decrease if patients do not maintain their physical activity level.

To change physical activity behaviour in is challenging. Different methods as Social Cognitive Theory, SCT and the Transtheoretical model, TTM have been suggested as theoretical framework. According to SCT, to improve physical activity behaviour you should use goal-setting, outcome expectancy, self-efficacy, and self-monitoring.

To use motivational interviewing (MI) improves the success of a behaviour change.

Patients will be randomized after the 12-week training period, tested, and thereafter both the intervention group and the control group will get information about the importance of physical activity and the recommendations.

Thereafter patients in the intervention group will receive weekly telephone calls for the first month, telephone calls every second week for the following two months and thereafter monthly telephone calls for the following three months. The telephone calls will be in accordance with MI and discuss goal-setting, out-come expectancy, and self-monitoring.

Patients will be tested after 6,12,and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD at Uppsala and Umeå university hospitals, who have participated in physical training at the hospital for 12 weeks.
* Diagnose of COPD

Exclusion criteria:

* Understand the Swedish language
* Be able to be physically active

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walking distance | Change from baseline and 6 months and up to 24 months
  Change in six-minute walking distance

SECONDARY OUTCOMES:
Physical activity level | Change from baseline and 6 months and up to 24 months
  Number of steps, energy expenditure, time in different positions
Short Form 36 | Change from baseline and 6 months and up to 24 months
  Measures health related quality of life
Chronic Respiratory Disease Questionnaire | Change from baseline and 6 months and up to 24 months
  Measures health related quality of life
Hospital anxiety and depression scale | Change from baseline and 6 months and up to 24 months
  Measures anxiety and depression
Grippit | Change from baseline and 6 months and up to 24 months
  Hand muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Emtner, PhD, Principal Investigator — Uppsala University; Karin Wadell, PhD, Study Chair — Umeå University
Locations (1):
- Uppsala University, Uppsala, Sweden